CLINICAL TRIAL: NCT01990599
Title: Airway Management in Patients Undergoing Thermal Ganglion Gasseri Coagulation, a New Method - Preliminary Results
Brief Title: Airway Management for Trigeminal Thermal Coagulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Wolfgang SCHRAMM, Univ. Prof. Dr., Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 1221/2012
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Airway Management
Keywords: nasopharyngeal tube; airway management; thermal coagulation of the Gasserian ganglion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nasopharyngeal Tube (Other): Every patient undergoing trigeminal thermal coagulation of the Gasserian ganglion will be ventilated by a nasopharyngeal placed ID 5mm tube during the whole neurosurgical intervention.
  Interventions: Other: Nasopharyngeal Tube

INTERVENTIONS:
Other: Nasopharyngeal Tube

SUMMARY:
Airway management of patients undergoing thermal coagulation of the Gasserian ganglion is very delicate. This is because of the specific operation site and moreover patients should recover quickly from anesthesia to follow verbal intraoperative commands of the surgeon. Endotracheal intubation or laryngeal mask of course hinders the patient from speaking. An obvious alternative airway management, as performed in this preliminary study, is a nasopharyngeal placed tube.

The purpose of the present study is to objectify the gas exchange in patients during this new ventilation technique.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing thermal coagulation of the Gasserian ganglion

Exclusion Criteria:

* Body weight over 100 kg
* Recurrent nasal bleeding
* Patients suffering from reflux disease
* Additional risk of aspiration (e.g. hernia diaphragmalis)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Blood gas exchange | Before and during the neurosurgical intervention
  Blood gas analyses will be determined at three time points perioperatively. The first measurement, at base line, will be performed preoperatively, the second one after puncture of the Gasserian ganglion and the third during the thermal coagulation of the Gasserian ganglion.

SECONDARY OUTCOMES:
SpO2 oxygen saturation (pulse oximeter) | Before and during the neurosurgical intervention
Hemodynamic parameters | Before and during the neurosurgical intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria